CLINICAL TRIAL: NCT02736994
Title: Assessment of the Impact of Probiotics on Biofilm Formation on Removable Acrylic Dentures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Supportive Care
Other Study IDs: S56279
Record Dates: First submitted 2014-01-17; First posted 2016-04-13 (Estimated); Last update posted 2016-04-13 (Estimated); Status verified 2013-11

CONDITIONS: Mandibular Prosthesis User
Keywords: edentulous; patients; with full
MeSH Terms: conditions — Mouth, Edentulous | interventions — Probiotics; Water

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Immersion in water (Other): water
  Interventions: Other: Water
- Immersion in water + cleansing tablet (Active Comparator): Corega Tabs Anti-bacteria® (GlaxoSmithKline Consumer Healthcare SA, Genval, Belgium)
  Interventions: Drug: Corega Tabs Anti-bacteria®
- Immersion in water with PIP (Experimental): PIP toothbrush cleaner® (Chrisal, Lommel, Belgium)
  Interventions: Drug: PIP toothbrush cleaner® (Chrisal, Lommel, Belgium).

INTERVENTIONS:
Drug: PIP toothbrush cleaner® (Chrisal, Lommel, Belgium). — Probiotic
  Other Names: Probiotic
  Arms: Immersion in water with PIP
Drug: Corega Tabs Anti-bacteria® — Cleansing tablet -Corega Tabs Anti-bacteria® (GlaxoSmithKline Consumer Healthcare SA, Genval, Belgium)
  Other Names: Cleansing tablet
  Arms: Immersion in water + cleansing tablet
Other: Water — Water
  Arms: Immersion in water

SUMMARY:
The aim of this study is to evaluate the effect of PIP toothbrush cleaner® on the microbial composition and Candida albicans colonization of denture biofilm formation. Additionally, its effect will be compared to that of cleansing tablets.

DETAILED DESCRIPTION:
Therefore the present study intended to compare a probiotic denture cleaning protocol with the current protocols. It was aimed to examine, in institutionalized older individuals with removable complete dentures, if the microbial composition and C. albicans colonization of the denture biofilm differs when overnight stored in a probiotic cleaning product compared to water or a cleanser. Additionally the influence of brushing on these protocols was investigated.

ELIGIBILITY:
Inclusion Criteria:

* Reside in a home for elderly
* Fully edentulous in lower and upper jaw
* Removable denture wearer in lower and upper jaw
* Good oral health

Exclusion Criteria:

* Current or history of corticosteroid treatment within the 3 months prior to the study
* Current or history of antimicrobial treatment within the 3 months prior to the study
* Inability to provide informed consent
* Inability to comply with the study requirements
* Heart disorders persons with a high risk for an unfavourable prognosis of bacterial endocarditis will be excluded. This applies to patients with prosthetic heart valves, history of infectious endocarditis, cyanogenic congenital heart disorders (including palliative shunts and connections), completely recovered congenital disorders that were treated less than 6 months ago, treated congenital heart disorders with residual defect, and valvulopathy after heart transplantation.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2014-04; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Candida albicans colonization | day 5
  C. albicans colonization was the primary outcome measure of interest. With a microbial test there was researched if C. albicans colonized the prostheses.

SECONDARY OUTCOMES:
Other microbiological counts Aa | day 5
  The concentration of Aggregatibacter Actinomycetemcomitans was researched.
Other microbiological counts Pg | day 5
  The concentration of Porphyromonas gingivalis was researched.
Other microbiological counts Tf | day 5
  The concentration of Tannerella forsythensis was researched.
Other microbiological counts Td | day 5
  The concentration of Treponema denticola was researched.
Other microbiological counts Pi | day 5
  The concentration of Prevotella intermedia was researched.
Other microbiological counts Fn | day 5
  The concentration of Fusobacterium nucleatum was researched.
Other microbiological counts Pm | day 5
  The concentration of Peptostreptococcus micros was researched.
Other microbiological counts Pn | day 5
  The concentration of Prevotella nigrescens was researched.
Other microbiological counts Cg | day 5
  The concentration of Campylobacter gracilis was researched.
Other microbiological counts Cr | day 5
  The concentration of Campylobacter rectus was researched.
Other microbiological counts En | day 5
  The concentration of Eubacterium nodatum was researched.
Other microbiological counts Ec | day 5
  The concentration of Eikenella corrodens was researched.
Other microbiological counts Capn | day 5
  The concentration of Capnocytophaga species was researched.
Other microbiological counts Cc | day 5
  The concentration of Campylobacter concisus count was researched.
Other microbiological counts mitis streptococci | day 5
  Concentration of mitis streptococci
Other microbiological counts Sg | day 5
  The concentration of Streptococcus gordonii
Other microbiological counts Sc | day 5
  The concentration of Streptococcus constellatus.
Other microbiological counts Ao | day 5
  The concentration of Actinomyces odontolyticus.
Other microbiological counts Av | day 5
  The concentration of Actinomyces viscosus.
Other microbiological counts Vp | day 5
  The concentration of Veillonella parvula.
Other microbiological counts total | day 5
  Total bacterial count.

CONTACTS AND LOCATIONS:
Overall Officials: Joke Duyck, DDS, PhD, Study Director — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- Department of Oral Health Sciences, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Duyck J, Vandamme K, Muller P, Teughels W. Overnight storage of removable dentures in alkaline peroxide-based tablets affects biofilm mass and composition. J Dent. 2013 Dec;41(12):1281-9. doi: 10.1016/j.jdent.2013.08.002. Epub 2013 Aug 13. PMID 23948391